CLINICAL TRIAL: NCT04939844
Title: Isatuximab in Combination With Bortezomib and Lenalidomide With Minimal Dexamethasone in Transplant-ineligible Multiple Myeloma
Brief Title: REST - Replacing Steroids in the Transplant Ineligble
Acronym: REST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Nordic Myeloma Study Group (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Fredrik Hellem Schjesvold, Head of Oslo Myeloma Center., Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMC02/20
Record Dates: First submitted 2021-04-07; First posted 2021-06-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Bortezomib; Lenalidomide

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, investigator initiated, single arm, open-label, multicenter study of isatuximab in combination with bortezomib and lenalidomide (IVR) with minimal dexamethasone, in patients with newly diagnosed multiple myeloma (NDMM) in-eligible for high dose melphalan with autologous stem cell support (HD-ASCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NDMM ineligible for transplant (Experimental): All participants will receive isatuximab in combination with bortezomib, lenalidomide and dexamethasone for 2 cycles, followed by isatuximab in combination with bortezomib and lenalidomide for 6 cycles, followed by isatuximab in combination with lenalidomide for 10 cycles, followed by continuous lenalidomide until disease progression. The cycle duration is 28 days.
  * Isatuximab will be administered IV at a dose of 10 mg/kg
    * on D1, D8, D15 and D22 during Cycle 1
    * on D1 and D15 during Cycles 2-18
  * Bortezomib will be administered SC at a dose of 1,3mg/m2
    -on D1, D8 and D15 during Cycles 1-8
  * Lenalidomide will be administered PO at a dose of 25mg/day (15 mg/day in participants with GFR <30mL/minute/1.73m2)
    -on D1 to D21 during all Cycles.
  * Dexamethasone will be administered PO at a dose of 20 mg -on D1, D8, D15 and D22 during Cycles 1 and 2
  Interventions: Drug: Isatuximab, bortezomib, lenalidomide, dexamethason

INTERVENTIONS:
Drug: Isatuximab, bortezomib, lenalidomide, dexamethason — All participants will receive the same treatment as described under arm.

SUMMARY:
Newly diagnosed multiple myeloma patients ineligible for HD-ASCT will be included in the study. All participants will receive isatuximab in combination with bortezomib, lenalidomide and minimal dexamethasone until disease progression. The primary objective of this study is the MRD negativity rate during and/or after first 18 cycles of study treatment.

DETAILED DESCRIPTION:
Approximately 53 participants will be screened to achieve 50 enrolled (sample size) to study intervention.All participants will receive isatuximab in combination with bortezomib, lenalidomide and dexamethasone for 2 cycles, followed by isatuximab in combination with bortezomib and lenalidomide for 6 cycles, followed by isatuximab in combination with lenalidomide for 10 cycles, followed by continuous lenalidomide until disease progression. The cycle duration is 28 days.Bone marrow MRD Euroflow NGF will be assessed once in participants achieving CR/sCR during the first 18 cycles of treatment, and in all participants (except for those who already are defined as MRD negative) achieving VGPR or better after finishing the first 18 cycles of treatment to assess. Those who are in VGPR and are MRD negative after 18 cycles of treatment will be response evaluated monthly for up to 4 months and if they become >CR during this period they are defined as MRD negative. The cut-off for MRD negativity is 100 plasma cells per 100 million nucleated cells (10-5).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Voluntary written informed consent.
2. Participant must be >18 years of age at the time of signing the informed consent.
3. Newly diagnosed multiple myeloma (IMWG criteria) in-eligible for high-dose therapy and ASCT.
4. Measurable disease as defined by the International Myeloma Working Group:

   1. Serum monoclonal paraprotein (M-protein) level > 10 g/L or urine M-protein level >200 mg/24 hours; or
   2. Light chain multiple myeloma without measurable disease in the serum or the urine: Involved serum immunoglobulin FLC > 100 mg/L and abnormal serum immunoglobulin kappa lambda FLC ratio.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2. ECOG 3 can only be enrolled if caused by myeloma.
6. Clinical laboratory values meeting the following criteria during the Screening Phase:

   a. Adequate bone marrow function:
   * Hemoglobin >7,5 g/dL (transfusion is permitted, recombinant human EPO use is permitted, however transfusion is not permitted within 3 days before screening)
   * Absolute neutrophil count > 1.0 x 109/L (G-CSF use is permitted)
   * Platelet count >70 x 109/L

     a) Adequate renal function:
   * eGFR>30 mL/min/m2
7. Patient must be willing and able to adhere to the study protocol visit schedule and other protocol requirements.
8. Females of childbearing potential (FCBPs) must have a confirmed negative serum or urine pregnancy test within 10-14 days prior to and again within 24 hours prior to starting study medication.
9. FCBPs and male subjects who are sexually active with FCBP must agree to use highly effective concomitant methods of contraceptive during the intervention period, for at least 5 months after last dose of isatuximab treatment and at least 28 days after last lenalidomide treatment. Male subjects must refrain from donating sperm during this period.

Exclusion Criteria:

1. Prior or current systemic therapy for multiple myeloma with the exception of emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
2. Radiation therapy for treatment of plasmacytoma(s) within 14 days before treatment (local radiation for pain control or to prevent fracture is allowed within 14 days before treatment).
3. Active hepatitis B or C virus infection or known human immunodeficiency virus (HIV) positivity.
4. Any other serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
5. No active malignancy with a lower life expectancy than myeloma.
6. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
7. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
MRD negativity | 34 months
  The proportion of patients who achieve MRD negativity measured by NGF Euroflow during and/or after 18 cycles of study treatment.

SECONDARY OUTCOMES:
Overall response rate | 30 months
  The proportion of patients who achieve partial response (PR) or better following 18 cycles of study treatment
Progression free survival | 4 years
  The PFS rate of patients receiving 2 cycles of IVRd followed by 6 cycles of IVR, 10 cycles of IR and continuous R
Overall survival | 5 years
  The OS rate of patients receiving 2 cycles of IVRd followed by 6 cycles of IVR, 10 cycles of IR and continuous R.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Schjesvold, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (4):
- Zealand University Hospital, Roskilde, Denmark
- Norway (3):
  - Oslo University Hospital, Oslo
  - Helse Stavanger HF, Stavanger
  - St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askeland FB, Haukas E, Slordahl TS, Klostergaard A, Alexandersen T, Lysen A, Abdollahi P, Nielsen LK, Hermansen E, Schjesvold F. Isatuximab, bortezomib, lenalidomide, and limited dexamethasone in patients with transplant-ineligible multiple myeloma (REST): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2025 Feb;12(2):e120-e127. doi: 10.1016/S2352-3026(24)00347-8. PMID 39909655